CLINICAL TRIAL: NCT02453880
Title: Web-based "Self-Help" Cognitive Behavioral Therapy for Symptoms of Mild-to-Moderate Anxiety and Depression in Adolescents and Young Adults With Chronic Illness
Brief Title: Web-based CBT for Symptoms of Mild-to-Moderate Anxiety and Depression in Youth With Chronic Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Rachel Bensen, MD, MPH, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 29456
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Depression; Anxiety; Inflammatory Bowel Disease; Systemic Lupus Erythematosus; Juvenile Idiopathic Arthritis
Keywords: anxiety; depression; chronic illness; teen; young adult
MeSH Terms: conditions — Depression; Anxiety Disorders; Inflammatory Bowel Diseases; Lupus Erythematosus, Systemic; Arthritis, Juvenile; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Web-based Cognitive Behavioral Therapy (Experimental): Participants will be directed to a web-based CBT "self-help" program with weekly modules.
  Interventions: Behavioral: Web-based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Web-based Cognitive Behavioral Therapy — Participants will be asked to complete a web-based cognitive behavioral therapy "self-help" program. The program consists of six weekly modules, in which participants practice new ways of thinking (e.g. how to recognize and change distorted thinking, utilizing a thought change record, identifying cognitive errors, and modifying automatic thoughts) to reduce symptoms of anxiety and depression. Participants receive text message reminders to complete the weekly session.

SUMMARY:
Symptoms of anxiety and depression are common in adolescents and young adults with chronic illnesses and are associated with decreased adherence to medical regimens. However, many young patients go untreated for anxiety and depression. The purpose of this study is to evaluate an online cognitive behavioral therapy (CBT) program in young adults with chronic illness. Prior research has shown online CBT to be effective in multiple other populations, but to the investigators' knowledge, this is the first study to examine web-based CBT for young adults with chronic illnesses.

DETAILED DESCRIPTION:
Emotional problems such as anxiety and depression commonly surface during adolescence and are even more common among youth with chronic illness compared to other children. Emotional comorbidities are associated with decreased adherence to medical regimens in children and adults as well as poorer clinical outcomes for medical conditions and increased medical expenditures. It is widely accepted that cognitive behavioral therapy is an effective treatment for anxiety and depression and in-person CBT has been shown effective for young people with inflammatory bowel disease (IBD). However, despite the presence of this effective treatment, the majority of those with anxiety and depression are untreated.

Offering mental health services in an acceptable, feasible and low cost fashion remains a challenge.

Research suggests that web-based CBT is a promising candidate for offering effective and feasible treatment for anxiety and depression to young people. It has been shown effective for mild to moderate symptoms of depression and anxiety in adults and adolescents with a primary diagnosis of depression. In adults, studies comparing face-to-face CBT treatment to web-based CBT with low level therapist support showed comparable clinical outcomes and a 15% cost savings for online treatment. Furthermore, an online treatment format may be especially appealing for younger populations who spend much of their time online as well as for people with chronic illness, who may be home-bound due to symptoms. Despite the well-established evidence base for web-based CBT in other populations, the greater affordability of web-based CBT compared to face-to-face treatment, and the appeal of the online format for young adults, the investigators are aware of no published studies examining the use of web-based CBT for young adults with chronic illness. The innovation of the proposed project is to study low- cost, web-based CBT in a new population of adolescents and young adults with inflammatory conditions that constitute serious chronic illness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic illness
* Language: English
* Computer and Internet access
* Symptoms of mild-moderate depression and/or anxiety

Exclusion Criteria:

* Existing mental health diagnosis
* Psychoactive medications initiated in past 2 months
* Severe depression
* Suicidal ideation (refer to on-call psychiatrist and/or social worker for urgent intervention) or history of prior suicide attempt

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Program completion rates | 6 weeks
  Intervention completion rates will be used as a marker for acceptability of the intervention.

SECONDARY OUTCOMES:
Change in pre-and post-intervention score on measure of depression (PHQ-9) | Baseline and 3 months
Change in pre-and post-intervention score on measure of anxiety (GAD-7) | Baseline and 3 months
Change in pre-and post-intervention score on measure of quality of life (Peds-QL) | Baseline and 3 months
Change in pre-and post-intervention score on measure of patient activation (PAM) | Baseline and 3 months

OTHER OUTCOMES:
Program satisfaction survey | 3 months
  Satisfaction with the web-based program will be assessed with a survey 3 months after enrollment in the study.